CLINICAL TRIAL: NCT04126876
Title: A Randomized Controlled Phase II Clinical Trial With Intradermal IMO-2125 (Tilsotolimod) in pT3-4 cN0M0 Melanoma
Brief Title: A Randomized Controlled Phase II Trial With Intradermal IMO-2125 in Pathological Tumor Stage (p) T3-4 cN0M0 Melanoma
Acronym: INTRIM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: A.J.M. van den Eertwegh (Other)
Collaborators: Idera Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, A.J.M. van den Eertwegh, Principal Investigator, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018/418
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — tilsotolimod; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Phase II Multicenter Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Persons that are masked/ blinded for which medication the patient receives: participant, treating physician/ team (including the person giving the intradermal injection) and peron who collects the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tilsotolimod (IMO-2125) (Experimental): Intradermal, single injection of 1 ml (8 mg) Tilsotolimod (IMO-2125) at the primary melanoma excision site, one week prior to sentinel node biopsy (SNB).
  Interventions: Drug: Tilsotolimod
- Placebo (Placebo Comparator): Intradermal, single injection of 1 ml plain saline (0.9% sodium chloride) at the primary melanoma excision site, one week prior to sentinel node biopsy (SNB).
  Interventions: Drug: Saline (0.9% sodium chloride)

INTERVENTIONS:
Drug: Tilsotolimod — Intradermal, single injection of 1 ml (8 mg) Tilsotolimod (IMO-2125) at the primary melanoma excision site, one week prior to sentinel node biopsy (SNB).
  Other Names: IMO-2125
  Arms: Tilsotolimod (IMO-2125)
Drug: Saline (0.9% sodium chloride) — Intradermal, single injection of 1 ml plain saline (0.9% sodium chloride) at the primary melanoma excision site, one week prior to sentinel node biopsy (SNB).
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Currently, there is no widely used adjuvant treatment available to improve survival after surgical excision of a primary melanoma. In a previous study, loco-regional and systemic immune stimulations, as well as favourable clinical outcomes in terms of sentinel lymph node (SLN) tumor status and recurrence-free survival (RFS) in patients with clinical stage I-II melanoma who received a low dose of toll-like receptor 9 (TLR-9) CPG7909 (CpG-B ODN) intradermally at the excision site of the primary tumor prior to SLN biopsy (SNB) were described. In this phase II trial the investigators had investigated the clinical activity of a next-generation CpG-ODN, IMO-2125, and it's ability to induce loco-regional and systemic immune stimulation in pT3-4 cN0M0 melanoma patients who are scheduled to undergo a combined re-excision and SNB is

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Histologically confirmed primary malignant melanoma cutis with a Breslow tumor depth >2.0 mm
* Scheduled to undergo a combines re-excision and sentinel node biopsy (SNB)
* World Health Organization (WHO) Performance Status ≤1
* Agreement to use effective contraceptive methods from screening until at least 90 days after the IMO-2125 administration
* Written informed consent

Exclusion Criteria:

* Known hypersensitivity to any oligodeoxynucleotide
* Active auto-immune disease requiring disease-modifying therapy at the tumr of screening
* Pathologically confirmed loco-regional or distant metastasis
* Non-skin melanoma
* Patients with another primary malignancy (some exceptions)
* Active systemic infections requiring antibiotics
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
The rate of tumor positive sentinal lymph node (SLN) | Seven days after the intradermal injection of Tilsotolimod (IMO-2125)
  The rate of tumor positive sentinal lymph node (SLN)

SECONDARY OUTCOMES:
Immune response in the SLN and peripheral blood | Seven days after the intradermal injection of Tilsotolimod (IMO-2125)
  Frequency and activation state of lymph node resident (LNR) conventional dendritic cells (DC) and melanoma antigen-specific T cell responses in the SLN and peripheral blood.
Recurrence free survival (RFS) | At 5 years and 10 years after sentinel node biopsy (SNB)
  The length of time from intradermal injection of Tilsotolimod (IMO-2125) to first documentation of recurrence.
Overall survival | At 5 years and 10 years after sentinel node biopsy (SNB)
  The length of time from intradermal injection of Tilsotolimod (IMO-2125) to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja de Gruijl, Principal Investigator — Amsterdam UMC, location VUmc; Alfons JM van den Eertwegh, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Centere, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koster BD, van den Hout MFCM, Sluijter BJR, Molenkamp BG, Vuylsteke RJCLM, Baars A, van Leeuwen PAM, Scheper RJ, Petrousjka van den Tol M, van den Eertwegh AJM, de Gruijl TD. Local Adjuvant Treatment with Low-Dose CpG-B Offers Durable Protection against Disease Recurrence in Clinical Stage I-II Melanoma: Data from Two Randomized Phase II Trials. Clin Cancer Res. 2017 Oct 1;23(19):5679-5686. doi: 10.1158/1078-0432.CCR-17-0944. PMID 28972083